CLINICAL TRIAL: NCT04195906
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of SNF472 When Added to Background Care for the Treatment of Calciphylaxis
Brief Title: Phase 3 Study of SNF472 for Calciphylaxis
Acronym: Calciphyx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanifit Therapeutics S. A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNFCT2017-06
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Calciphylaxis; Calcific Uremic Arteriolopathy
Keywords: Calciphylaxis; Calcific Uremic Arteriolopathy; Wound; ESRD
MeSH Terms: conditions — Calciphylaxis; Wounds and Injuries; Kidney Failure, Chronic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SNF472 (Double-Blind Period) (Experimental): Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline.
  Interventions: Drug: Experimental: SNF472
- Placebo (Double-Blind Period) (Placebo Comparator): Matching placebo (saline) diluted in 100 mL physiological saline.
  Interventions: Drug: Placebo Comparator: Placebo
- SNF472 (Open-Label) (Experimental): Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline.
  Interventions: Drug: Experimatenl SNF472 (Open-label)

INTERVENTIONS:
Drug: Experimental: SNF472 — Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks
  Arms: SNF472 (Double-Blind Period)
Drug: Placebo Comparator: Placebo — Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions fo 12 weeks
  Other Names: Saline
  Arms: Placebo (Double-Blind Period)
Drug: Experimatenl SNF472 (Open-label) — Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks
  Arms: SNF472 (Open-Label)

SUMMARY:
The primary objectives are to assess the efficacy, safety, and tolerability of SNF472 compared to placebo when added to background care for the treatment of calciphylaxis (CUA).

DETAILED DESCRIPTION:
The formation and growth of calcified deposits in arterioles and other small blood vessels appears to be fundamental to the development of CUA especially in end stage renal disease patients. This phase 3 double-blind, randomized, placebo-controlled study is designed to assess the effect of SNF472 when added to background care to improve wound healing, as evaluated using Bates-Jensen Wound Assessment Tool (BWAT) scoring and pain as reported by the subject using a VAS scale. The study consists of a double-blind, randomized, placebo controlled period of 12 weeks followed by an open-label period of 12 weeks.. .

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects, 18 years of age or older
* Receiving maintenance HD in a clinical setting for at least 2 weeks prior to screening
* Clinical diagnosis of CUA by the Investigator including ≥1 CUA lesion with ulceration of the epithelial surface
* CUA wound-related pain shown by a Pain VAS score ≥50 out of 100
* Primary lesion that can be clearly photographed for the purpose of protocol-specified wound healing assessments.
* Willing and able to understand and sign the informed consent form and willing to comply with all aspects of the protocol

Exclusion Criteria:

* History of treatment with bisphosphonates within 3 months of baseline
* Severely ill subjects without a reasonable expectation of survival for at least 6 months
* Subjects with a scheduled parathyroidectomy during the study period
* Expectation for kidney transplant within the next 6 months based on Investigator assessment or identification of a known living donor
* Pregnant or trying to become pregnant, currently breastfeeding, or of childbearing potential (including perimenopausal women who have had a menstrual period within one year) and not willing to comply with protocol required contraception criteria
* Significant noncompliance with dialysis
* History of active malignancy within the last year with the exception of localized basal cell or squamous cell carcinoma
* Clinically significant illness other than CUA within 30 days
* Participation in an investigational study and receipt of an investigational drug or investigational use of a licensed drug within 30 days prior to screening.
* History or presence of active alcoholism or drug abuse as determined by the Investigator within 6 months
* Mental impairment, current significant psychiatric disease, or other conditions or circumstances that would make the subject unlikely to complete the study or comply with the study procedures.
* Subjects whose CUA lesions exhibit significant improvement, in the opinion of the Investigator, between the first and second screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Gold, MD, Study Director — Sanifit Therapeutics
Locations (58):
- United States (38):
  - AKDHC Medical Research Services, Phoenix, Arizona
  - California Institute of Renal Research, El Centro, California
  - California Institute of Renal Research, Escondido, California
  - Kidney Disease Medical Group, Glendale, California
  - DaVita Clinical Research, Lynwood, California
  - Apex Research of Riverside, Riverside, California
  - Fresenius Kidney Care, San Diego, California
  - North America Research Institute, San Dimas, California
  - Amicis Research Center, Vacaville, California
  - Colorado Kidney Care, Denver, Colorado
  - Boca Nephrology, PA, Boca Raton, Florida
  - DaVita Clinical Research, Hollywood, Florida
  - Novel Outcomes Research, Spring Hill, Florida
  - DaVita Clinical Research, Tampa, Florida
  - Fresenius Kidney Care, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Kidney Consultants, Pontiac, Michigan
  - DaVita Clinical Research, Roseville, Michigan
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Fresenius Kidney Care, Brookhaven, Mississippi
  - DaVita Clinical Research, Kansas City, Missouri
  - DaVita Clinical Research, Las Vegas, Nevada
  - Fresenius Kidney Care, Reno, Nevada
  - DaVita Clinical Research, The Bronx, New York
  - DaVita Clinical Research, Asheville, North Carolina
  - Fresenius Kidney Care, Durham, North Carolina
  - Piedmont Dialysis Center, Winston-Salem, North Carolina
  - Hypertension Nephrology Consultants, Inc, Columbus, Ohio
  - Fresenius Kidney Care, Bethlehem, Pennsylvania
  - DaVita Clinical Research, Chester, Pennsylvania
  - Fresenius Kidney Care, Columbia, South Carolina
  - Knoxville Kidney Center, Knoxville, Tennessee
  - DaVita Clinical Research, Houston, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - DaVita Clinical Research, Chesapeake, Virginia
  - DaVita Clinical Research, Norfolk, Virginia
  - Fresenius Kidney Care, Roanoke, Virginia
  - DaVita Clinical Research, Wauwatosa, Wisconsin
- Belgium (3):
  - Clinques Universitaries de Bruxelles Hopital, Brussels
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
- Germany (3):
  - Nephrologischen Zentrum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - DaVita Deutschland AG, Düsseldorf
- Poland (5):
  - Centrum Dializ Fresenius, Ośrodek Dializ nr 10 w Bydgoszczy 85-826, Bydgoszcz
  - Centrum Dializ Fresenius, Ośrodek Dializ nr 18 w Krakowie.., Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego w Lodzi Stacja Dializ,, Lodz
  - DaVita Sp. z o.o., Stacja Dializ w Miechowie, Miechów
  - Centrum Dializ Fresenius Ośrodek Dializ nr 32 w Radomiu 26-617 ., Radom
- Spain (3):
  - Fundacio Puigvert, Barcelona
  - University of Barcelona Hospital Clinic, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
- United Kingdom (6):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Leicester General Hospital, Leicester, Leicestershire
  - Queen Elizabeth University Hospital Campus, Glasgow, Strathclyde
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinha S, Nigwekar SU, Brandenburg V, Gould LJ, Serena TE, Moe SM, Aronoff GR, Chatoth DK, Hymes JL, Carroll KJ, Alperovich G, Keller LH, Perello J, Gold A, Chertow GM. Hexasodium fytate for the treatment of calciphylaxis: a randomised, double-blind, phase 3, placebo-controlled trial with an open-label extension. EClinicalMedicine. 2024 Aug 16;75:102784. doi: 10.1016/j.eclinm.2024.102784. eCollection 2024 Sep. PMID 39252867
- [Derived] Krishnasamy R, Jardine MJ; BEAT-Calci Trialists. Adaptive Designs for Clinical Trials in Nephrology. J Am Soc Nephrol. 2025 Jan 1;36(1):147-149. doi: 10.1681/ASN.0000000000000497. Epub 2024 Aug 26. No abstract available. PMID 39186385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 148 participants were screened in 48 sites in 5 countries; 77 participants were not enrolled because they were screen failures (did not meet eligibility criteria). A total of 71 participants were randomized in the study to receive SNF472 or placebo.
Groups:
- SNF472 (Double-blind Period + Open-label): Part 1 (double-blind period):
  Participants received SNF472 for 12 weeks in addition to their background care.
  Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
  Part 2 (Open-label):
  Participants received SNF472 for 12 weeks in addition to their background care.
  Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
- Placebo (Double-blind Period) + SNF472 (Open-label): Part 1 (double-blind period) Participants received placebo for 12 weeks in addition to their background care.
  Dose: Matching placebo (saline) diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions fo 12 weeks
  Part 2 (Open-label):
  Participants received SNF472 for 12 weeks in addition to their background care.
  Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
Period: Part 1
Arm/Group | SNF472 (Double-blind Period + Open-label) | Placebo (Double-blind Period) + SNF472 (Open-label)
Started | 37 | 34
Completed | 34 | 26
Not Completed | 3 | 8
Not completed — Adverse Event | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1
Period: Part 2
Arm/Group | SNF472 (Double-blind Period + Open-label) | Placebo (Double-blind Period) + SNF472 (Open-label)
Started | 34 | 26
Completed | 32 | 19
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat Population (mITT): The modified mITT population was defined as all enrolled subjects who were randomized, received at least one dose of study drug, and had at least one post-randomization efficacy evaluation.
  The mITT population was the primary analysis population for efficacy endpoints.
Groups:
- SNF472: Part 1 (double-blind period):
  Participants received SNF472 for 12 weeks in addition to their background care. Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
  Part 2 (Open-label):
  Participants received SNF472 for 12 weeks in addition to their background care. Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
- Placebo: Part 1 (double-blind period) Participants received placebo for 12 weeks in addition to their background care.
  Dose: Matching placebo (saline) diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions fo 12 weeks.
  Part 2 (Open-label):
  Participants received SNF472 for 12 weeks in addition to their background care. Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline. Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | SNF472 | Placebo | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.14) | 57.2 (11.30) | 57.5 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 14 | 12 | 26
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Europe | 5 | 2 | 7
  North America | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the BWAT - CUA Score for the Primary Lesion
Description: The Bates Jensen Wound Assessment Tool (BWAT) CUA score ranges from a minimum score of 8 (best) to a maximum score of 40 (worst).
  BWAT-CUA= Bates-Jensen Wound Assessment Tool-Calcific Uremic Arteriolopathy
Time Frame: from Baseline to Week 12
Population: Modified Intent-to-treat Population (mITT) population: defined as all enrolled subjects who were randomized, received at least one dose of study drug, and had at least one post-randomization efficacy evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SNF472: Participants who received SNF472 for 12 weeks in addition to their background care during the double-blind period (Part 1).
  Dose: 7 mg/kg SNF472 diluted in 100 mL physiological saline.
  Experimental: SNF472: Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions for 12 weeks
- Placebo: Participants who received placebo for 12 weeks in addition to their background care during the double-blind period (Part 1).
  Matching placebo (saline) diluted in 100 mL physiological saline.
  Placebo Comparator: Placebo: Administered 3 times weekly by intravenous infusion through the hemodialysis machine in conjunction with the subject's hemodialysis sessions fo 12 weeks
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
score on a scale | -5.3 (5.18) | -6.0 (6.17)
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.877, MMRM — The MMRM model includes fixed effect terms for randomized treatment, visit, baseline sodium thiosulfate use, baseline BWAT-CUA score and visit by randomized treatment interaction; MMRM=Mixed model for repeated measures Participant is fitted as random effect and an unstructured variance-covariance matrix is used; Least Squares Mean Difference = 0.27, 96% CI 2-sided [-2.46 to 3.00], Standard Error of Mean 1.328

2. Primary Outcome: Absolute Change in Pain Visual Analog Score
Description: The Pain Visual Analog Scale (VAS) score ranges from a minimum score of 0 (no pain) to 100 (worst possible pain).
Time Frame: from Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
score on a scale | -19.5 (26.89) | -32.2 (38.53)
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.146, MMRM — The MMRM model includes fixed effect terms for randomized treatment, visit, baseline sodium thiosulfate use, baseline Pain VAS and visit by randomized treatment interaction; MMRM: mixed model repeated measures. Participant is fitted as random effect and an unstructured variance-covariance matrix is used; Least Squares Mean Difference = 11.49, 96% CI 2-sided [-4.80 to 27.78], Standard Error of Mean 7.930

3. Secondary Outcome: Absolute Change in the Wound-Quality of Life Score
Description: The Wound Quality of Life scale is a validated self-assessment tool that has been shown to be feasible for assessing health-related quality of life in patients with chronic wounds. Lower scores are associated with a better quality of life as reported by the patient.
  The score is computed by averaging the 17 items on impairments assessed on a scale of 0 to 4 for the preceding 7 days. A global score can only be computed if at least 75% of the items have been answered, i.e., at least 13 in 17 items are valid. All the available items' scores were added up and divided by 17. In case of missing assessments for any one of the 17 items, the median of the scores for a particular item within the associated randomized treatment group was used for the imputation purposes.
  As the absolute change from baseline is reported, a higher negative value is associated with a higher improvement of quality of life.
Time Frame: from Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
score on a scale | -0.67 (0.798) | -0.74 (1.175)
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.706, MMRM — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.09, 96% CI 2-sided [-0.38 to 0.56], Standard Error of Mean 0.237

4. Secondary Outcome: Absolute Change in the BWAT Total Score for the Primary Lesion
Description: The Bates Jensen Wound Assessment Tool (BWAT) score ranges from a minimum score of 9 (best) to a maximum score of 65 (worst) score.
Time Frame: from Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
score on a scale | -11.0 (9.85) | -11.7 (12.23)
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.995, MMRM — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.02, 96% CI 2-sided [-5.27 to 5.24], Standard Error of Mean 2.630

5. Secondary Outcome: Qualitative Wound Image Evaluation for the Primary Lesion
Description: A qualitative assessment (Worsened, Equal to, or Improved Relative to Baseline) was assigned
Time Frame: at Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
Participants
  Worsened | 6 | 7
  Equal | 0 | 1
  Improved | 23 | 18
  Missing | 8 | 8
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.384, Regression, Logistic — This model includes the stratification factor sodium thiosulfate use at baseline and the treatment as covariates; As there is only a measure post-baseline, a logistic regression model was run instead of a generalized estimating equations model; Odds Ratio, log = 1.54, 95% CI 2-sided [0.58 to 4.09], Standard Error of Mean 0.498 — The odds ratio displayed is the odds ratio of having an improved result of SNF472 versus Placebo. The results 'Worsened', 'Equal', and 'Missing' are combined in one category and it is the reference for the odds ratio calculation

6. Secondary Outcome: Rate of Change in Opioid Use as Measured in Morphine Milligram Equivalents (MME)
Description: Change from baseline in opioid use MME = Morphine Milligram Equivalents
  The calculation of the pre-specified list of opioids was based on the formula: strength per unit × (number of units/days supply) × MME conversion factor = MME/day, as specified in the opioid MME conversion guide (CMS, 2017). The maintenance opioid dose was defined as the average daily opioid dose in MME during the 7-day period prior to Screening Visit 2.
  To assess the extent to which opioid use may have differed between randomized treatment groups over time, the change from baseline in daily average MME value was analyzed.
Time Frame: from Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: MME/week
Arm/Group | SNF472 | Placebo
Number analyzed (Participants) | 37 | 34
MME/week | 0.46 (0.461) | -0.11 (0.499)
Statistical Analysis 1: Comparison: SNF472 vs Placebo; Test type: Superiority; p = 0.406, MMRM — MMRM model includes fixed effect terms for randomized treatment, continuous variables maintenance opioid dose, Week (1 to 12) and Week by randomized treatment interaction. The random coefficients are the intercept and Week as a continuous variable; MMRM: mixed model repeated measures. An unstructured variance-covariance matrix is used; Difference in slopes between arms = 0.57, 95% CI 2-sided [-0.79 to 1.93], Standard Error of Mean 0.680

ADVERSE EVENTS:
Time Frame: Part 1: 12-week double-blind, randomized, placebo-controlled treatment period Part 2: 12-week open-label treatment period after completion of part 1 period.
Groups:
- SNF472 - Safety Analysis Population (Part 1): Participants who received SNF472 treatment during part 1 (Double-blind Period).
  The number of participants in the safety set differs from the previous figures provided in the Participant Flow section, as 1 participant associated to placebo arm, by mistake, actually received a few infusions with SNF472. As a consequence, this participant is counted within the SNF472 Safety Analysis Population (making it 38 subjects instead of 37).
- Placebo - Safety Analysis Population (Part 1): Participants who received placebo during part 1 (Double-blind Period).
- SNF472 Open Label - Safety Analysis Population (Part 2): Participants who received SNF472 treatment during part 2 (Open-label)
Arm/Group | SNF472 - Safety Analysis Population (Part 1) | Placebo - Safety Analysis Population (Part 1) | SNF472 Open Label - Safety Analysis Population (Part 2)
All-Cause Mortality (participants affected / at risk) | 1/38 | 6/33 | 1/60
Serious Adverse Events (participants affected / at risk) | 13/38 | 17/33 | 18/60
Other Adverse Events (participants affected / at risk) | 27/38 | 21/33 | 33/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 - Safety Analysis Population (Part 1) (N=38) | Placebo - Safety Analysis Population (Part 1) (N=33) | SNF472 Open Label - Safety Analysis Population (Part 2) (N=60)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNF472 - Safety Analysis Population (Part 1) (N=38) | Placebo - Safety Analysis Population (Part 1) (N=33) | SNF472 Open Label - Safety Analysis Population (Part 2) (N=60)
Calciphylaxis (Metabolism and nutrition disorders) | 8 (9) | 8 (9) | 4 (8)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 3 (3) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (2) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 2 (5) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Hypervolemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04195906/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT04195906/SAP_001.pdf